CLINICAL TRIAL: NCT07230288
Title: A Phase 2a Multicenter Platform Study of Investigational Products for the Treatment of Adult Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Study of ABBV-142 to Assess Adverse Events and Change in Disease Activity in Adult Participants With Idiopathic Pulmonary Fibrosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M25-268; 2024-518013-25-00 (Other: EU CT)
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Substudy 1: ABBV-142 (Experimental): Participants will receive ABBV-142 for 52 week during double-blind treatment period. Eligible participants may receive ABBV-142 for 52 weeks during open-label treatment period.
  Interventions: Drug: ABBV-142
- Substudy 1: Placebo for ABBV-142 (Placebo Comparator): Participants will receive placebo for ABBV-142 for 52 week during double-blind treatment period. Eligible participants may receive ABBV-142 for 52 weeks during open-label treatment period.
  Interventions: Drug: ABBV-142; Drug: Placebo for ABBV-142

INTERVENTIONS:
Drug: ABBV-142 — ABBV-142
Drug: Placebo for ABBV-142 — Placebo for ABBV-142
  Arms: Substudy 1: Placebo for ABBV-142

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a rare, long-lasting lung disease that causes scarring of lung tissue, shortness of breath, and loss of lung function. IPF leads to significant loss of quality of life and shortened lifespan. This study is a platform study evaluating different types of treatments in patients with IPF. A platform study is a type of study that uses a single master protocol to evaluate different study treatments allowing for new study treatments or substudies to be added or closed over time. The main goals of the study are to evaluate the safety, tolerability (the degree to which the adverse symptoms can be handled by the patients during the study) and efficacy (how well study treatment works) of the study treatments, including ABBV-142 in Substudy 1 (SS1).

ABBV-142 is an investigational drug being developed for the treatment of IPF. In SS1, participants will be randomly assigned to one of the 2 groups to receive either ABBV-142 or a matching placebo. This study is "double-blind", meaning that neither the participants nor the study doctors know who is given which study treatment. Approximately 165 adult participants with IPF will be enrolled in approximately 125 sites across the world.

Participants will receive ABBV-142 or matching placebo for 52 weeks during the double-blind treatment period. Eligible participants may receive ABBV-142 for 52 weeks in open-label treatment period. All participants will be followed for 120 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of Idiopathic Pulmonary Fibrosis (IPF) within 7 years prior to screening, confirmed by the investigator at screening that is supported by centrally read chest high-resolution computed tomography (HRCT) obtained within 12 months of the screening visit and verification of usual interstitial pneumonia(UIP) or probable UIP.

Exclusion Criteria:

* History of stroke within 6 months prior to screening
* In the opinion of the investigator, other clinically significant pulmonary abnormalities
* History of any malignancy up to 5 years prior screening visit, except for successfully treated nonmelanoma skin cancer or localized carcinoma in situ of the cervix.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Absolute Change From Baseline in Forced Vital Capacity (FVC) (mL) | Week 24
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Percentage of Participants with Adverse Events (AE) | Up to approximately 52 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Absolute Change From Baseline in Forced Vital Capacity (FVC) (mL) | Week 52
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Relative Change From Baseline in FVC (mL) | Week 24
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Relative Change From Baseline in FVC (ml) | Week 52
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Absolute Change from Baseline in FVC% predicted | Up to approximately 52 weeks
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Relative Change From Baseline in FVC% predicted | Up to approximately 52 weeks
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Change From Baseline in Living with Pulmonary Fibrosis (L-PF) Overall Score | Up to approximately 52 weeks
  L-PF questionnaire is a 49-item disease specific PRO that assesses symptoms and impacts of living with pulmonary fibrosis among participants with fibrosing interstitial lung disease (ILD). Summary scores range from 0-100, the higher the score the greater the impairment.
Time to First Absolute Decline From Baseline in FVC% Predicted of >= 10% | Up to approximately 52 weeks
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Time to First Relative Decline From Baseline in FVC% Predicted of >= 10% | Up to approximately 52 weeks
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Time to First Absolute Decline From Baseline in FVC% Predicted >= 5% | Up to approximately 52 weeks
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.
Time to First Relative Decline From Baseline in FVC% Predicted >= 5% | Up to approximately 52 weeks
  FVC is a test that measures the total amount of air a person can fully exhale from their lungs after a deep inhalation. A low FVC can demonstrate reduced lung capacity.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-268